CLINICAL TRIAL: NCT00642200
Title: Lichtenstein Hernioplasty Versus Totally Extraperitoneal Laparoscopic Hernioplasty in Treatment of Recurrent Inguinal Hernia - A Prospective Randomized Trial
Brief Title: Recurrent Inguinal Hernia Treatment - Lichtenstein Versus Laparoscopic Totally Extraperitoneal Preperitoneal Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Collaborators: University of Kuopio Computing Center (Unknown)
Responsible Party: MD Sanna Kouhia, North Karelia Central Hospital, Clinic of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKCH-surg-001
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Recurrent Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients receive Lichtenstein hernioplasty as a treatment for recurrent inguinal hernia.
  Interventions: Procedure: Lichtenstein hernioplasty
- 2 (Active Comparator): Patients receive laparoscopic TEP as a treatment for recurrent inguinal hernia.
  Interventions: Procedure: Laparoscopic TEP

INTERVENTIONS:
Procedure: Lichtenstein hernioplasty
  Arms: 1
Procedure: Laparoscopic TEP
  Arms: 2

SUMMARY:
The study aims at detecting possible differences between an open (Lichtenstein) and a video-assisted (TEP) technique in treating recurrent inguinal hernia. The differences monitored are further recurrence and chronic pain as well as primary complications.

ELIGIBILITY:
Inclusion Criteria:

* recurrent inguinal hernia
* willing to participate

Exclusion Criteria:

* unwilling to participate
* bilateral hernia
* preference towards either treatment arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1997-01; Primary Completion 2002-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
further recurrence | 3 weeks, 1 year, 2 years, 3 years

SECONDARY OUTCOMES:
chronic pain or discomfort | 3 weeks, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- North Karelia Central Hospital - Clinic of Surgery, Joensuu, Pohjois-Karjala, Finland

REFERENCES:
- [Derived] Kouhia ST, Huttunen R, Silvasti SO, Heiskanen JT, Ahtola H, Uotila-Nieminen M, Kiviniemi VV, Hakala T. Lichtenstein hernioplasty versus totally extraperitoneal laparoscopic hernioplasty in treatment of recurrent inguinal hernia--a prospective randomized trial. Ann Surg. 2009 Mar;249(3):384-7. doi: 10.1097/SLA.0b013e318196d0b0. PMID 19247022